CLINICAL TRIAL: NCT04512118
Title: CT Abnormalities Evocative of Lung Infection Are Associated With Lower 18F-FDG Uptake in Confirmed COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, PhD, Central Hospital, Nancy, France
Other Study IDs: 2020PI153
Record Dates: First submitted 2020-08-12; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Presence of COVID-19 Compatible CT Abnormalities
Keywords: COVID19; 18F FDG PET; lung infection; CT; seriological tests
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET-CT of 18F-FDG — Whole-body 18F-FDG-PET/CT was performed on a digital hybrid system (Vereos, Philips®)

SUMMARY:
CT signs that are evocative of lung COVID-19 infections have been extensively described, whereas 18F-FDG-PET signs have not. Our current study aimed to identify specific COVID-19 18F-FDG-PET signs in patients that were (i) suspected to have a lung infection based on 18F-FDG-PET/CT recorded during the COVID-19 outbreak and (ii) whose COVID-19 diagnosis was definitely established or excluded by appropriate viral testing.

ELIGIBILITY:
Inclusion Criteria:

* Patient coming to nuclear medicine for 18F-flurodesoxyglucose (FDG) positron emission tomography computed tomography (PET-CT) with suspicion of lung involvement
* patient affiliated to a social security scheme or equivalent
* adult patient having been informed of the study

Exclusion Criteria:

* patient with a negative covid 19 test

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with suspicion of lung involvement in COVID19 context
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Visual analysis of pulmonary lobes | 1 day
  Visual analysis of the pulmonary lobes by calculating a extent score for each patient

SECONDARY OUTCOMES:
Measurement of metabolic activity | 1 day
  Measurement of metabolic activity with SUV max of lung areas with CT abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU of Nancy, Vandœuvre-lès-Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: No